CLINICAL TRIAL: NCT04030676
Title: Place of the QuantiFERON-CMV (QF-CMV) Test in a Prediction for Colic Cytomegalovirus Reactivation During Ulcerative Colitis (UC)
Brief Title: QuantiFERON-CMV Test in a Prediction for Colic Cytomegalovirus Reactivation During Ulcerative Colitis
Acronym: RECOHFERRON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18CH053; 2018-A01622-53 (Other: ANSM)
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cytomegalovirus Infections
Keywords: Immune response against; QuantiFERON-CytoMegaloVirus (QF-CMV); Ulcerative Colitis (UC); CytoMegaloVirus (CMV); quantitative PolymeraseChainReaction (qPCR); ImmunoHistoChemistry (IHC)
MeSH Terms: conditions — Cytomegalovirus Infections; Colitis, Ulcerative | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QuantiFERON Test (Experimental): Patient with CytoMegaloVirus (CMV) infection will be included. They will have biopsies and blood samples, composite of QuantiFERON-CytoMegaloVirus (QF-CMV) assay.
  Interventions: Procedure: Biopsies; Biological: Blood samples

INTERVENTIONS:
Procedure: Biopsies — Two more biopsies in inflammatory zone will be collected.
Biological: Blood samples — Blood samples will be performed necessary at QuantiFERON-CMV (QF-CMV) test.

SUMMARY:
CytoMegaloVirus (CMV) infection impairs evolution of Ulcerative Colitis (UC) leading to more severe and resistant to immunosuppressive therapies flare-up. CytoMegaloVirus (CMV) reactivation is assessed by the quantification of the CytoMegaloVirus (CMV) DeoxyriboNucleic Acid (DNA) load by real-time PCR (qPCR) in colonic biopsies; this assay is invasive and costly. The QuantiFERON-CytoMegaloVirus (QF-CMV) assay measures the immune response against CytoMegaloVirus (CMV) in a blood specimen.

DETAILED DESCRIPTION:
This study aim to evaluate the performances of this new assay to predict the risk of CytoMegaloVirus (CMV) reactivation in the colon of UC patients. A new algorithm for the care of Ulcerative Colitis (UC) patients that could be used in all centers, even those without molecular biology lab, could be proposed: in case of a positive QuantiFERON-CytoMegaloVirus (QF-CMV) assay, the immune response protects the patient against Cytomegalovirus (CMV) reactivation and intensification of immunosuppressive therapies should be proposed; at the opposite, a negative QuantiFERON-CytoMegaloVirus (QF-CMV) assay will invite to biopsy in order to detect CytoMegaloVirus (CMV) replication and to treat with ganciclovir when appropriate. This algorithm will preserve invasive biopsies in absence of CytoMegaloVirus (CMV) tissue reactivation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with seropositive for CytoMegaloVirus (CMV) (IgG+)
* Patient requiring hospitalization for flare of Ulcerative Colitis (UC) with Mayo score > 5 and an endoscopic subscore ≥ 2
* Social security affiliation
* Signed informed consent

Exclusion Criteria:

* Wardship patient and curatorial patient
* Patient unable to understand or sign the protocol
* Colectomy total or partial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Quantification of CytoMegaloVirus (CMV) DeoxyriboNucleic Acid (DNA) load (quantitative PolymeraseChainReaction (qPCR) analysis) in the inflammatory tissue - UI/100 000 cells | At the inclusion
  Theses two primary outcomes will determinate the sensibility, specificity, positive predictive value and negative predictive value of the QF-CMV in prediction CMV reactivation in Ulcerative Colitis (UC) patients with acute flare-up.
QuantiFERON-CytoMegaloVirus (QF-CMV) test result (UI/ml) in blood | At the inclusion
  Theses two primary outcomes will determinate the sensibility, specificity, positive predictive value and negative predictive value of the QF-CMV in prediction CMV reactivation in Ulcerative Colitis (UC) patients with acute flare-up.

SECONDARY OUTCOMES:
Total number of cells infected by CMV (/mm2) by ImmunoHistoChemistry (IHC) in the inflammatory tissue | At the inclusion
  To determine the performance threshold of the QuantiFERON-CytoMegaloVirus (QF-CMV) assay as assessed by ImmunoHistoChemistry (IHC) that can predict CytoMegaloVirus (CMV) reactivation in colonic biopsies in Ulcerative Colitis (UC) patients with acute flare-up.
Concordance of the results between quantitative PolymeraseChainReaction (qPCR) and ImmunoHistoChemistry (IHC) | At the inclusion
  To evaluate the concordance of the results between quantitative PolymeraseChainReaction (qPCR) and ImmunoHistoChemistry (IHC) analysis.
QuantiFERON-CytoMegaloVirus (QF-CMV) test result (UI/ml) in blood | At 14 weeks
  To compare measure of the QuantiFERON-CytoMegaloVirus (QF-CMV) assay at the flare-up and 14 weeks after.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ROBLIN, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Sylvie PILLET, PhD, Study Director — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - HCL-Hôpital Lyon Sud, Lyon
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No